CLINICAL TRIAL: NCT02268266
Title: ERIGO® Life - Study of Cardiovascular Parameters and Other Physiologic Parameters Under Verticalization and Simultaneous Mobilization of the Leg on Neurological Patients and Healthy Subjects
Brief Title: ERIGO® Life- Control of Cardiovascular Parameters Via Verticalization and Simultaneous Mobilization
Acronym: ERIGO®LIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Zuercher Hoehenklinik Wald (Other); Hocoma AG, Switzerland (Unknown)
Responsible Party: Principal Investigator, Verena Klamroth, Dr. med., Swiss Federal Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERIGO LIFE StV 22_2009
Record Dates: First submitted 2014-07-31; First posted 2014-10-20 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Stroke; Spinal Cord Injury
Keywords: brain injury, early rehabilitation, tilt table
MeSH Terms: conditions — Stroke; Spinal Cord Injuries; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm study (Other): Early mobilization of patients after stroke or spinal cord injury. Monitoring of vital parameters during mobilization of healthy subjects
  Interventions: Device: Erigo

INTERVENTIONS:
Device: Erigo — The control of cardiovascular parameters within suitable ranges for healthy and neurological patients using verticalization, leg mobilization and electrical stimulation
  Other Names: Erigo rehabilitation bed from Hocoma AG, Switzerland.

SUMMARY:
Early verticalization and stepping with the equipment of Hocoma ERIGO during monitoring of vital parameters. The device is already CE marked and, for the purposes of the study, will be used in accordance with the intended use (after-market clinical investigation).

DETAILED DESCRIPTION:
In early rehabilitation of neurological patients, safe mobilization and intensive sensorimotor stimulation are key factors for therapeutic success. Early activation and stimulation of the patient intend enhancement of neuroplasticity and recovery. Furthermore, it improves the patient's communication and cooperation skills and counteracts secondary damages due to immobilization.

The study combines gradual verticalization during monitoring of vital parameters, with cyclic leg movement and foot loading. The table to ensures the necessary safety for the stabilization of the patient in the upright position. The patient stimulation is additionally enhanced by synchronized functional electrical stimulation (FES). By providing a safe solution for early mobilization, the Erigo counteracts the negative effects of immobility and accelerates the recovery process through intensive sensorimotor stimulation. It is the first choice therapy device for the early and safe mobilization of severely impaired, bed-ridden patients even in acute care.

ELIGIBILITY:
Inclusion criteria:

* minimum 18 years old
* normal response to verbal instructions
* oxygen saturation of the blood at least 92%
* healthy german speaking men and women
* non-smoker
* heartbeat 40-100
* systolic blood pressure 120 to 220 mmHg
* in patients: post acute phase: stroke or other neurological functional disorder

Exclusion criteria:

* severe contraction in the legs (Ashworth >3)
* pregnancy
* acute pain syndrome
* severe cardio-pulmonary disease
* history of orthostatic dysregulation
* thrombophlebitis
* diabetes
* renal disease
* contraindication for electric stimulation (instable epilepsy, cancer, pacemaker, palliative care)
* weight > 120kg
* height > 210 cm
* skin lesions on legs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse event as a measure of safety and tolerability | Up to 8 hours
  Control of cardiovascular parameters at desired ranges at healthy and at patients

CONTACTS AND LOCATIONS:
Overall Officials: Robert Riener, Prof.Dr.-Ing, Principal Investigator — Swiss Federal Institut of Technology
Locations (2):
- Switzerland (2):
  - Zürcher Höhenklinik Wald, Wald, Canton of Zurich
  - ETH Zurich, Zurich, Canton of Zurich